CLINICAL TRIAL: NCT06586502
Title: Responding to Late Effects in Survivors of Childhood Cancer (RECOVER)
Brief Title: Responding to Late Effects in Survivors of Childhood Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Remziye Semerci (Other)
Responsible Party: Sponsor-Investigator, Remziye Semerci, Associate Professor, Trakya University
Organization: Trakya University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: QUT
Record Dates: First submitted 2024-08-19; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Survivorship; Model of Care; Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): We will compare outcomes of a historical control group, matched for child age and diagnosis, as closely as possible to identify any significant differences between groups that may be attributed to the RECOVER Model of care.
- Intervention Group (Experimental): The intervention group in the RECOVER study consists of cancer survivors aged 15-39 years who have completed treatment, along with their carers or parents, and health professionals. The survivors will undergo a comprehensive health assessment, including both physical and psychological aspects, to inform the development of a personalized care plan. Carers or parents, who must be able to read and understand English or work with an interpreter, will be actively involved in the assessment process and subsequent consultations to help shape the care plan. Health professionals, including doctors, nurses, and allied health providers from Queensland Health public hospitals, will participate in multidisciplinary team meetings, review health assessments, and contribute to the creation and implementation of the care plan. These groups together form the core of the intervention, engaging in both the application and evaluation of the RECOVER Model of Car
  Interventions: Other: Model of Care

INTERVENTIONS:
Other: Model of Care — The intervention described in the RECOVER study involves developing, implementing, and evaluating a comprehensive Model of Care for childhood cancer survivors. This model, known as the RECOVER Model of Care, integrates digital health solutions and is co-designed with input from childhood cancer survivors, caregivers, and clinical experts. The intervention aims to address the long-term and late effects of cancer treatment by providing continuous, risk-based, interdisciplinary care. It includes steps such as identifying patients nearing the end of treatment, conducting health assessments, creating personalized care plans, and coordinating follow-up care through digital platforms. The study will assess the feasibility, acceptability, and effectiveness of this model in improving the quality of life and care experience for survivors and their families.
  Arms: Intervention Group

SUMMARY:
Survivors of childhood cancer need ongoing support to navigate their needs after cancer treatment. Using technology may offer us new ways to collect and share information about cancer survivorship follow-up with young survivors, their carers, and primary care providers.

Through the support of the Kids Cancer Project, in Phase 1 of this study, will co-design an electronic survivorship 'portal' that links young survivors with their cancer treatment information, and health care teams. In later Phases we will implement and evaluate the survivorship portal.

DETAILED DESCRIPTION:
The RECOVER study aims to develop and implement a comprehensive Model of Care for childhood cancer survivors, integrating technology and a human-centered co-design approach to provide continuous, holistic care. Our primary objectives are to assess the feasibility and acceptability of the RECOVER Model of Care in routine pediatric oncology practice. Secondary objectives include evaluating preliminary efficacy results and identifying factors that influence the successful adoption and integration of the model.

Data Sources: This project will be conducted in three settings in Australia. The study will use a mixed methods approach, starting with a feasibility study (Phase 1), following implementation science methods to assess the integration of the new Model of Care (Phase 2), and culminating in a Type 2 Hybrid Implementation/Effectiveness non-randomized controlled trial (Phase 3) to compare historical and prospective data. The quantitative component of RECOVER (non-randomized controlled study) will involve the use of digital technologies to (1) enable multimodal, real-world data collection, (2) provide patients and caregivers with an interactive, supportive digital interface, and (3) equip healthcare professionals with a comprehensive patient-monitoring system. The qualitative component will determine end-user feasibility and acceptability through focus group workshops, surveys, and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15-39 years who have completed cancer treatment.
* Ability to read and understand English.
* Willingness to comply with study procedures and provide informed consent.
* Clinicians (doctors, nurses, allied health professionals) providing care through *Queensland Health public hospitals

Exclusion Criteria:

* Patients deemed unsuitable by their clinical treatment team due to potential distress or lack of cognitive or communicative capacity.
* None specified, as long as they meet the inclusion criteria.

Max Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Caregiver Quality of Life Cancer | Baseline, Sixth and twelfth month
  The scale is a validated and reliable measure, comprising 35 items on a 5-point Likert scale, which we have widely used in other studies with this population (Weitzner et al., 1999). We will compare outcomes of a historical control group (N=100), matched for child age and diagnosis, as closely as possible to identify any significant differences between groups that may be attributed to the RECOVER Model of care.
Pediatric Integrated Care Survey | Baseline, Sixth and twelfth month
  Pediatric Integrated Care Survey
Distress Thermometer for Parents | Baseline, Sixth and twelfth month
  The DT-P is a valid and reliable short screening tool for identifying parental distress. It was developed to determine parents' distress who had chronically ill children (0-18 years). The DT-P consists of a thermometer score from 0 (no distress) to 10 (extreme distress) and a problem list (practical, social, emotional, physical, cognitive, and parenting domains) (Haverman et al., 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bradford, Bradford, Principal Investigator — Cancer and Palliative Care Outcomes Centre
Locations (1):
- Queensland Children's Hospital, Brisbane, Center, Australia

IPD SHARING:
Plan to Share IPD: No